CLINICAL TRIAL: NCT03501927
Title: The Effects of Pre-operative Point-of-Care Focused Cardiac Ultrasound on Patient Outcome - a Prospective, Randomized, Clinical Study (PreOPFOCUS)
Brief Title: Focused Cardiac Ultrasound in Surgery
Acronym: PreOPFOCUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossible patient inclusion due to the COVID-10 pandemic
Sponsor: Aarhus University Hospital (Other)
Collaborators: Randers Regional Hospital (Other); Aabenraa Hospital (Other)
Responsible Party: Principal Investigator, Jan Pallesen, Principal Investigator, Randers Regional Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PreOPFOCUS
Record Dates: First submitted 2018-02-20; First posted 2018-04-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cardiopulmonary Disease; Surgery; Morality; Complication
Keywords: Ultrasound; FOCUS; Surgery; Anesthesia
MeSH Terms: conditions — Pulmonary Heart Disease

STUDY DESIGN:
Intervention Model Description: Preoperative point-of-care focused cardiopulmonary ultrasound (FOCUS) Patients are to be randomised in a 1:1 ratio to either 1) FOCUS prior to anaesthesia or 2) no FOCUS performed (standard treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOCUS (focused cardiac ultrasound) (Active Comparator): Patients allocated to FOCUS will receive a preoperative FOCUS examination in conjunction with a standard anesthetic preoperative evaluation.
  Interventions: Diagnostic Test: FOCUS (focused cardiac ultrasound)
- Control (No Intervention): Patients allocated til control arm will receive a standard anesthetic preoperative evaluation according to hospitals' standards.

INTERVENTIONS:
Diagnostic Test: FOCUS (focused cardiac ultrasound) — A ultrasound of the heart and pleura will be performed. This provide information on
  * Left ventricular systolic function
  * Left ventricular diastolic function
  * Right ventricular systolic function
  * Right ventricular pressure overload
  * Biventricular sizes
  * Pathology of the mitral- and aortic valves
  * Pericardial fluid
  * Gross fluid status
  * Pleural effusion
  Arms: FOCUS (focused cardiac ultrasound)

SUMMARY:
Mortality and morbidity remain high after non-cardiac surgery. Known risk factors include age, high ASA grade and emergency surgery. Point-of-care focused cardiac ultrasound may elucidate pathology and potential hemodynamic compromise unknown to handling physicians. This study aims to investigate the effects of focused cardiac ultrasound in high-risk patients undergoing non-cardiac surgery with respect to clinical endpoints.

DETAILED DESCRIPTION:
In non-cardiac surgery major risk factors for morbidity and mortality include ASA classification, age, acute surgery and pre-existing cardiopulmonary disease. These risk factors are sometimes readily available and, along with the type of surgery, allow anaesthesiologists to tailor anaesthetic drugs, fluid therapy and monitoring to the individual patient need. However, cardiopulmonary disease may be occult or masked by other patient-related incapacities. Hence, identification of cardiopulmonary disease is an important priority during the pre-operative anaesthesia evaluation. Routine pre-operative anaesthesia evaluation includes screening with auscultation, blood tests and often electrocardiography. However, these exams are insensitive for detecting cardiopulmonary diseases that may be life threatening during anaesthesia, including ischaemia, heart valve disease and left ventricular hypertrophy.

Point-of-care focused cardiac ultrasound (FOCUS) is claimed to be an effective method for filling out this obvious gap in rapid diagnostic capability, as FOCUS can detect both structural and functional cardiac disease as well as pleural effusion. FOCUS performed by anaesthesiologists can identify unknown pathologies in surgical patients and identification of these enables prediction of perioperative morbidity. Although pre-operative FOCUS has been shown to alter anaesthetic patient management, it remains unclear whether the application of FOCUS actually impacts patient outcome.

This study aims to clarify whether pre-operative FOCUS changes clinical outcomes in high-risk patients undergoing acute, non-cardiac surgery.

The hypothesis of the study is that pre-operative FOCUS reduces the fraction of patients admitted to hospital for more than 10 days or are dead within 30 days after high risk, non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for emergency (< 6 hours) or urgent surgery (< 24 hours)15
* General or neuro-axial anaesthesia planned at the first anesthetic visit
* ASA classification 3 or 4.
* Age ≥ 65 years

Exclusion Criteria:

* Previous surgery performed during current hospital admission (including transfers from other hospitals than Randers Regional Hospital/Hospital of Southern Jutland)
* Low risk surgery or expected surgery time < 30 minutes or endoscopies.
* Lack of consent from patient or proxy (in case of patient mental incapacity)
* Previous participation in the study. Pre-operative FOCUS not possible for logistical reasons or due to requirement for immediate surgery

Drop-out Criteria:

Patients who refuse participation after formal inclusion will drop out.

• Patients converted from a primary anaesthetic plan of general/neuro-axial anaesthesia to regional anaesthesia will not drop-out. -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 337 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients admitted to hospital ≥ 10 days or dead within 30 days | 30 days after surgery

SECONDARY OUTCOMES:
Length of stay | Up to 180 days after surgery
  Defined as the number of days admitted to hospital from the date of surgery (included)
Re-admissions to hospital | Up to 90 days after surgery
  Re-admissions to hospital (no) within 90 days (no)
Length of stay | Up to 90 days after surgery
  Length of stay including re-admissions to hospital within 90 days
Death ≤ 30 days & ≤ 90 days | Up to 90 days after surgery
  Death ≤ 30 days & ≤ 90 days (no)
Intensive care treatment | Up to 90 days after surgery
  Intensive care treatment (hours)
Postoperative ventilator treatment | Up to 90 days after surgery
  Postoperative ventilator treatment (hours)
Admittance to the post-operative care unit | Up to 1 day after surgery
  Admittance to the post-operative care unit (hours)
Development of acute kidney injury | Within 7 days of surgery
  Development of acute kidney injury (AKI) (stage 1,2 & 3, defined by th KDIGO creatinine criteria within seven days of surgery)
Accumulated intra- and postoperative infusion of norepinephrine, epinephrine, phenylephrine, ephedrine, dobutamine, dopamine and other vasoactive drugs. | From start of anaesthesia til end of anaesthesia
  Accumulated intra- and postoperative infusion of norepinephrine, epinephrine, phenylephrine, ephedrine, dobutamine, dopamine and other vasoactive drugs (mg).
Accumulated fluid balance | From start of anaesthesia til end of anaesthesia
  Accumulated fluid balance until end of surgery
Echocardiography | From anaeshetic visit to start of anaesthesia
  Formal echocardiography's (1) ordered and (2) actually performed in total and secondarily due to preoperative FOCUS (no).
Surgery cancellations due to preoperative FOCUS | Before start of anaeshesia
  Surgery cancellations in total and secondarily due to preoperative FOCUS (no)
Surgery postponements due to preoperative FOCUS | Within 7 days of preoperative anaesthetic visit
  Surgery postponements in total and secondarily due to preoperative FOCUS (no).
Surgery changes | From FOCUS to the start of surgery
  Surgery changes in total and secondarily due to preoperative FOCUS (no, type).
Perioperative myocardial damage | From the day before surgery to the day following surgery
  Troponin I
Changes in anesthetic practice | From start of anaesthesia to start of surgery
  Changes in anesthetic practice/perianesthetic care DUE to preoperative FOCUS. Includes both step up/step down
Echocardiography | From FOCUS to start of surgery
  Formal echocardiographies ordered prior to surgery
Volume | From FOCUS to the start of anaesthesia
  Volume infusion prior to anesthesia. Both in total and facilitated by FOCUS
Anaesthesia type | From FOCUS to the start of anaesthesia
  Conversion of Anaesthesia type from primary anesthetic visit to actually performed. Both in total and facilitated by FOCUS.
Anaesthetic monitoring | From start of anaesthesia to end of anaesthesia
  Step up and step down in anesthetic monitoring. Both in total and facilitated by FOCUS. Includes extra intravenous lines inserted including central venous catheters, arterial lines inserted, change to 5-lead ECG, vasopressors infused with anaesthetic induction
Anesthesia time | From start of anaesthesia to end of anaesthesia
  Anesthesia time
Surgery time | From start of surgery to end of surgery
  Surgery time
Cardiogenic pulmonary oedema | From start of anaesthesia to 30 days after surgery
  Cardiogenic pulmonary oedema within 30 days of surgery
New onset cardiac arrhythmia | From start of anaesthesia to 30 days after surgery
  New onset cardiac arrhythmia of any kind.
Non-fatal cardiac arrest | From start of anaesthesia to 30 days after surgery
  Non-fatal cardiac arrest regardless of cause.
Anastomotic breakdown | From start of anaesthesia to 30 days after surgery
  Anastomotic breakdown (deep or superficial)
Myocardial infarction | From start of anaesthesia to 30 days after surgery
  Myocardial infarction as defined by the universal criteria
Stroke | From start of anaesthesia to 30 days after surgery
  Cerebral stroke
Pulmonary embolism | From start of anaesthesia to 30 days after surgery
  Pulmonary embolism with radiological confirmation
Postoperative haemorrhage | From end of anaesthesia to 30 days after surgery
  Postoperative haemorrhage demanding blood transfusion
Gastrointestinal bleed | From start of anaesthesia to 30 days after surgery
  Gastrointestinal bleed
Pneumonia | From start of anaesthesia to 30 days after surgery
  Pneumonia
Surgical site infection | From end of anaesthesia to 30 days after surgery
  Surgical site infection (superficial or deep)
Urinary tract infection | From end of anaesthesia to 30 days after surgery
  Urinary tract infection
Infektion, source unknown | From end of anaesthesia to 30 days after surgery
  Infektion, source unknown.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pallesen, MD, Principal Investigator — Randers Regional Hospital; Rajesh Bhavsar, MD, Principal Investigator — Aabenraa Hospital
Locations (1):
- Department of Anaesthesiology, Randers, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Protocol and statistical plan will be published in a peer-reviewed journal. Study results will be made available at a freely accessible online site.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol within 6 months of study commencement Study results within 6 months of study termination
Access Criteria: Public
URL: http://www.preopfocus.dk

REFERENCES:
- [Background] M Saklad. Grading patients for surgical procedures. Anesthesiology 1941;2:281-4
- [Background] Davenport DL, Ferraris VA, Hosokawa P, Henderson WG, Khuri SF, Mentzer RM Jr. Multivariable predictors of postoperative cardiac adverse events after general and vascular surgery: results from the patient safety in surgery study. J Am Coll Surg. 2007 Jun;204(6):1199-210. doi: 10.1016/j.jamcollsurg.2007.02.065. PMID 17544078
- [Background] Kheterpal S, O'Reilly M, Englesbe MJ, Rosenberg AL, Shanks AM, Zhang L, Rothman ED, Campbell DA, Tremper KK. Preoperative and intraoperative predictors of cardiac adverse events after general, vascular, and urological surgery. Anesthesiology. 2009 Jan;110(1):58-66. doi: 10.1097/ALN.0b013e318190b6dc. PMID 19104171
- [Background] Khuri SF, Henderson WG, DePalma RG, Mosca C, Healey NA, Kumbhani DJ; Participants in the VA National Surgical Quality Improvement Program. Determinants of long-term survival after major surgery and the adverse effect of postoperative complications. Ann Surg. 2005 Sep;242(3):326-41; discussion 341-3. doi: 10.1097/01.sla.0000179621.33268.83. PMID 16135919
- [Background] Asch FM, Shah S, Rattin C, Swaminathan S, Fuisz A, Lindsay J. Lack of sensitivity of the electrocardiogram for detection of old myocardial infarction: a cardiac magnetic resonance imaging study. Am Heart J. 2006 Oct;152(4):742-8. doi: 10.1016/j.ahj.2006.02.037. PMID 16996851
- [Background] Olive KE, Grassman ED. Mitral valve prolapse: comparison of diagnosis by physical examination and echocardiography. South Med J. 1990 Nov;83(11):1266-9. doi: 10.1097/00007611-199011000-00008. PMID 2237552
- [Background] Beyerbacht HP, Bax JJ, Lamb HJ, van der Laarse A, Vliegen HW, de Roos A, Zwinderman AH, van der Wall EE. Evaluation of ECG criteria for left ventricular hypertrophy before and after aortic valve replacement using magnetic resonance imaging. J Cardiovasc Magn Reson. 2003 Jul;5(3):465-74. doi: 10.1081/jcmr-120022262. PMID 12882077
- [Background] Holm JH, Frederiksen CA, Juhl-Olsen P, Sloth E. Perioperative use of focus assessed transthoracic echocardiography (FATE). Anesth Analg. 2012 Nov;115(5):1029-32. doi: 10.1213/ANE.0b013e31826dd867. Epub 2012 Oct 9. No abstract available. PMID 23051882
- [Background] Botker MT, Vang ML, Grofte T, Sloth E, Frederiksen CA. Routine pre-operative focused ultrasonography by anesthesiologists in patients undergoing urgent surgical procedures. Acta Anaesthesiol Scand. 2014 Aug;58(7):807-14. doi: 10.1111/aas.12343. Epub 2014 May 28. PMID 24865842
- [Background] Kratz T, Campo Dell'Orto M, Exner M, Timmesfeld N, Zoremba M, Wulf H, Steinfeldt T. Focused intraoperative transthoracic echocardiography by anesthesiologists: a feasibility study. Minerva Anestesiol. 2015 May;81(5):490-6. Epub 2014 Sep 15. PMID 25220551
- [Background] Cowie B. Focused transthoracic echocardiography predicts perioperative cardiovascular morbidity. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):989-93. doi: 10.1053/j.jvca.2012.06.031. Epub 2012 Aug 22. PMID 22920841
- [Background] Canty DJ, Royse CF, Kilpatrick D, Williams DL, Royse AG. The impact of pre-operative focused transthoracic echocardiography in emergency non-cardiac surgery patients with known or risk of cardiac disease. Anaesthesia. 2012 Jul;67(7):714-20. doi: 10.1111/j.1365-2044.2012.07118.x. Epub 2012 Mar 27. PMID 22452367
- [Background] Kratz T, Steinfeldt T, Exner M, Dell Orto MC, Timmesfeld N, Kratz C, Skrodzki M, Wulf H, Zoremba M. Impact of Focused Intraoperative Transthoracic Echocardiography by Anesthesiologists on Management in Hemodynamically Unstable High-Risk Noncardiac Surgery Patients. J Cardiothorac Vasc Anesth. 2017 Apr;31(2):602-609. doi: 10.1053/j.jvca.2016.11.002. Epub 2016 Nov 2. PMID 28089598
- [Background] Moore CL. Does Ultrasound Improve Clinical Outcomes? Prove It. Crit Care Med. 2015 Dec;43(12):2682-3. doi: 10.1097/CCM.0000000000001325. No abstract available. PMID 26575658
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN; American College of Cardiology; American Heart Association. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. J Am Coll Cardiol. 2014 Dec 9;64(22):e77-137. doi: 10.1016/j.jacc.2014.07.944. Epub 2014 Aug 1. No abstract available. PMID 25091544
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, Ford I, Gonzalez-Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luscher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Sousa-Uva M, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014 Sep 14;35(35):2383-431. doi: 10.1093/eurheartj/ehu282. Epub 2014 Aug 1. No abstract available. PMID 25086026
- [Background] Glance LG, Lustik SJ, Hannan EL, Osler TM, Mukamel DB, Qian F, Dick AW. The Surgical Mortality Probability Model: derivation and validation of a simple risk prediction rule for noncardiac surgery. Ann Surg. 2012 Apr;255(4):696-702. doi: 10.1097/SLA.0b013e31824b45af. PMID 22418007
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Background] Bilimoria KY, Liu Y, Paruch JL, Zhou L, Kmiecik TE, Ko CY, Cohen ME. Development and evaluation of the universal ACS NSQIP surgical risk calculator: a decision aid and informed consent tool for patients and surgeons. J Am Coll Surg. 2013 Nov;217(5):833-42.e1-3. doi: 10.1016/j.jamcollsurg.2013.07.385. Epub 2013 Sep 18. PMID 24055383
- [Background] Section 2: AKI Definition. Kidney Int Suppl (2011). 2012 Mar;2(1):19-36. doi: 10.1038/kisup.2011.32. No abstract available. PMID 25018918
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Tsang TS, Barnes ME, Gersh BJ, Bailey KR, Seward JB. Left atrial volume as a morphophysiologic expression of left ventricular diastolic dysfunction and relation to cardiovascular risk burden. Am J Cardiol. 2002 Dec 15;90(12):1284-9. doi: 10.1016/s0002-9149(02)02864-3. PMID 12480035
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Ryan T, Petrovic O, Dillon JC, Feigenbaum H, Conley MJ, Armstrong WF. An echocardiographic index for separation of right ventricular volume and pressure overload. J Am Coll Cardiol. 1985 Apr;5(4):918-27. doi: 10.1016/s0735-1097(85)80433-2. PMID 3973294
- [Background] Balik M, Plasil P, Waldauf P, Pazout J, Fric M, Otahal M, Pachl J. Ultrasound estimation of volume of pleural fluid in mechanically ventilated patients. Intensive Care Med. 2006 Feb;32(2):318. doi: 10.1007/s00134-005-0024-2. Epub 2006 Jan 24. PMID 16432674
- [Derived] Pallesen J, Bhavsar R, Fjolner J, Krog J, Malachauskiene L, Bakke SA, Andersen MAS, Vang ML, Andersen JK, Bondergaard MH, Jessing TD, Thee C, Mortensen L, Nielsen MB, Juhl-Olsen P. The effects of preoperative point-of-care focused cardiac ultrasound in high-risk patients: study protocol for a prospective randomised controlled trial. Dan Med J. 2020 Jan;67(1):A07190410. PMID 31908251